CLINICAL TRIAL: NCT05697133
Title: The Effect of Symptom Management Program Based on Story Theory on Vasomotor Symptoms and Sleep Quality in Postmenopausal Women
Brief Title: Symptom Management Program Based on Story Theory for Postmenopausal Women (SEMSTOP)
Acronym: SEMSTOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Emel Guven, Research Assistant, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21063324
Record Dates: First submitted 2022-11-30; First posted 2023-01-25 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Menopause
Keywords: Sleep Quality; Postmenopause
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEMSTOP (Experimental): It is the group to which the initiatives will be applied.
  Interventions: Other: SEMSTOP
- Control (Active Comparator): It is the group to be compared to which the interventions will not be applied.
  Interventions: Other: control

INTERVENTIONS:
Other: SEMSTOP — This program has been developed based on Story Theory and will be implemented individually online. The session content, units and topics in the program are arranged according to the conceptual content and flow of the theory. The program has been created in a certain flow, based on the concepts of purposeful dialogue, connecting with itself and facilitating the theory.
  Arms: SEMSTOP
Other: control — control grup
  Arms: Control

SUMMARY:
Purpose: To investigate the effect of the Symptom Management Program Based on Story Theory on vasomotor symptoms and sleep quality in postmenopausal women.

Design: The type of this research is mixed method (qualitative and quantitative research design together). It enables to strengthen the weaknesses of mixed method research, to increase the generalizability of the results, and to produce more reliable outputs regarding theory and practice. The quantitative research dimension is a randomized single-blind pretest-posttest experimental model with a control group. The qualitative research dimension is the descriptive phenomenological design.

Method: The research will be carried out at Ömürevleri, Atakum, Mimar Sinan, Çobanlı and Yenimahalle Family Health Centers located in different regions of the Atakum District of Samsun. After informing the women who come to the Family Health Centers about the face-to-face research, the research will be conducted completely online (due to the COVID-19 pandemic) after the verbal consent of the women who volunteered to participate in the research and their contact numbers are obtained. The postmenopausal women who apply to the institutions where the research will be conducted and meet the inclusion criteria constitute the population of the research. When the sample size calculated with the G.Power program was taken as Pittsburgh Sleep Quality Index score mean and standard deviation value as 6.57±1.23, with 5% significance level, 80% test power, 0.700 effect size, there were at least 68 groups, 34 for the experimental group and 34 for the control group. identified as a person. Considering the sample loss in the experimental and control groups, with 10% more sampling, a total of 76 women will be included in the sample, with 38 women in each group. n the study, the data will be collected with the Personal Information Form, the Menopause Symptoms Assessment Scale, the Pittsburgh Sleep Quality Index and the Story Theory Based Semi-Structured Interview Form (for qualitative research) developed by the researchers in line with the literature. As a result of the study, the data will be evaluated separately as qualitative and quantitative.

ELIGIBILITY:
Inclusion Criteria:

* Be a volunteer,
* To be literate to have a smart mobile phone/computer
* To be in the first 2 years after menopause
* Experiencing vasomotor symptoms

Exclusion Criteria:

* Having a communication barrier
* Having problems with internet access
* Being in the premenopausal period
* Undergoing surgical menopause
* Getting a diagnosis of respiratory system
* Getting a diagnosis of hypertension and cardiovascular disease
* Getting treatment for menopause, getting training on breathing exercises
* Treatment for sleep disorders receive

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index | 1st months
  It will be used to measure sleep qualıty of postmenoposal women
Menopause Symptoms Rating Scale | 1st months
  It will be used to evaluate menopaus symptoms of postmenoposal women

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index | 3rd months
  It will be used to measure sleep quality of postmenoposal women
Menopause Symptoms Rating Scale: | 3rd months
  It will be used to evaluate menopaus symptoms of postmenoposal women

IPD SHARING:
Plan to Share IPD: No